CLINICAL TRIAL: NCT03967899
Title: Study of Electrical Prognostic Factors of Response to Intravenous Immunoglobulin Treatment in Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: PRONELEC PIDC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRONELEC
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuropathy (PIDC) is an acquired dysimmune polyneuropathy whose prevalence is estimated to be between 1 to 4 per 100,000 depending on the study, with an incidence of less than 1 per 100,000 per year. The clinical presentation of PIDC is heterogeneous, characterized by a symmetrical lesion predominating generally on large fibers, the most myelinated, responsible for ataxia and a motor deficit in the foreground. In the typical form, patients describe a proximal and distal motor or sensory deficit associated with isflexia that signifies a peripheral neurogenic syndrome.

The physiopathological hypothesis is that of an inflammation responsible for demyelinating nerve fibers, which results in electroneuromyogram (ENMG) by conduction abnormalities and histologically when a neuromuscular biopsy is performed by segmental demyelination.

Given the heterogeneity of the clinical presentation, electrical diagnostic criteria are proposed by the European Federation of Neurological Society in order to classify IPDCs into three categories: certain, probable and possible. In the absence of sufficient criteria to make the diagnosis of IPDC, it is also possible to use criteria of support, using a paraclinical report including the presence of an increase in protein (hyperproteinorachie) without cells for cerebrospinal fluid analysis, visualization of radicular inflammation on imaging (MRI of lumbar and / or brachial plexus), proximal peripheral involvement with somatosensory evoked potentials.

Therapeutically, a joint management between rehabilitation and the introduction of a background treatment allows the clinical improvement of certain patients. To date, the treatments proposed in first intention are corticosteroids, intravenous immunoglobulins (IVIg) and plasma exchanges. In fact, the efficacy of intravenous immunoglobulins has been widely shown by controlled and randomized therapeutic trials. Efficacy studies of IVIg in the literature are most often based on an assessment of clinical response after 24 weeks, but in clinical practice the response to treatment and continuation of treatment is often evaluated after 3 courses of treatment with the help of a clinical evaluation and the realization of an electroneuromyogram. These are administered in day hospitalization or traditional hospitalization, every four weeks, to patients whose diagnosis of PIDC has been established by electroneuromyogram according to the EFNS criteria.

Clinical prognostic factors for good response to IVIG therapy have been described in previous studies, including subacute disease, symmetrical involvement, and absence of amyotrophy.

In order to optimize the management of IPDCs, it is important to identify patients who respond to IVIg. Thus, the objective of our study is to look at the electroneuromyogram, the presence of electrical predictors of good response to treatment with IVIg.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is ≥ 18 years
* Patients with IPDC
* Patients hospitalized in a traditional hospital ward or week hospital or day hospital
* Patients who received at least 3 courses of IVIG under IPDC between January 2014 and March 2019
* Francophone patients

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients who oppose the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPDC, hospitalized in a traditional hospital ward or week hospital or day hospital, who received at least 3 courses of IVIG under IPDC between January 2014 and March 2019
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Identify electromyographic predictors of treatment response | Week 24
  This corresponds to highlight, in the data of the electroneuromyogram performed before the initiation of treatment with IVIg, differences between the responder groups or not treatment [decrease of at least 1 point in the ONLS score], i.e three courses of IVIG.

SECONDARY OUTCOMES:
study of the demographic characteristics of patients followed for IPDC and treated with IVIg | Week 24
  This corresponds to percentage of patients with a certain / probable or possible IPDC.
Clinical evidence of response to IVIG treatment | Week 24
  comparison of the results of the complementary explorations in the patients answering or not to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pauline REACH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France